CLINICAL TRIAL: NCT06555991
Title: Translation and Validation of the Shoulder Instability Return to Sports Index (SIRSI) and Tampa Scale of Kinesiophobia Shoulder Instability (TSK-SI) Into German
Brief Title: Translation and Validation of the SIRSI and TSK-SI Into German
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Schulthess Klinik (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: OE-236
Record Dates: First submitted 2024-08-06; First posted 2024-08-15 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Shoulder Instability
Keywords: Return to Sports; Shoulder Instability; SIRSI; TSK-SI; Kinesiophobia
MeSH Terms: conditions — Kinesiophobia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SIRSI and TSK-SI (Other): The SIRSI and TSK-SI as well as the WOSI and RTS-, Clinical- and Demographic Information are gathered. The SIRSI and TSK-SI are re-administered one week later
  Interventions: Other: SIRSI and TSK-SI

INTERVENTIONS:
Other: SIRSI and TSK-SI — The SIRSI and TSK-SI as well as the WOSI and RTS-, Clinical- and Demographic Information are gathered. The SIRSI and TSK-SI are re-administered one week later

SUMMARY:
Clinicians need to evaluate the psychological readiness to return to sports after an shoulder injury. The SIRSI is a questionnaire that provides such information, however it has not yet been translated and tested for a German speaking population (Switzerland, Austria or Germany). Similarily the TSK-SI is a questionnaire that measures fear of movement in patients with shoulderinstability, which is also not available to German speaking patients.

This study is conducted to translate both questionnaires into German and test it in German speaking patients in Switzerland.

DETAILED DESCRIPTION:
Return to Sports (RTS) is an important outcome measure after shoulder instability treatment (Abdul-Rassoul et al., 2019). While the definition of returning to sport is not clear (Doege et al., 2021), efforts have been made to provide consensus. The concept of Return to Sport is multifactorial consisting of physical, psychological, and social/contextual factors in an interplay with sociodemographic and injury factors. Furthermore, different stages of RTS have been defined (Ardern et al., 2016). To take all factors into account, outcome measures like the ACL-RSI for anterior cruciate ligament ruptures have been invented (Webster et al., 2008). To provide such a measure for the shoulder instability cohort Gerometta et al (2018) have adapted the ACL-RSI to a shoulder instability population and named it the Shoulder Instability Return to Sport Index (SIRSI). Since then, this outcome has been frequently used to determine psychological readiness to RTS (Rossi et al., 2022). Despite an available German translation, published by a German insurance company (Return-to-Competition Schulter: Shoulder Instability-Return to Sport after Injury (SIRSI)-Skala (vbg.de), accessed 23.01.2024), the SIRSI is not scientifically available for a German speaking population, because this version has never been officially translated and validated. Similarly the Tampa Scale for Kinesiophobia (TSK) has been invented to measure an excessive fear of movement due to painful injury in chronic low back pain (Miller et al., 1991). The Scale was then adapted to the shoulder instability cohort (van Iersel et al., 2023). However, it is currently not available in German. Therefore, this project seeks to translate the SIRSI and TSK-SI into a German version and validate them in a German speaking population in Switzerland.

The aim of the project is to translate the Shoulder Instability Return to Sports Index (SIRSI) and Tampa Scale for Kinesiophobia - Shoulder Instability (TSK-SI) into a German version and assess its validity in a Swiss-German population of patients with shoulder instability treated conservatively or surgically and planning to return to sports.

ELIGIBILITY:
Inclusion Criteria:

1. Had an instability event within last year
2. Provided general consent for local shoulder instability register at Schulthess Klinik Zürich
3. Adult patients aged 18 or older

Exclusion Criteria:

1. Are at least three months after surgery or instability event
2. Must endeavor to return to their sport
3. Have another physical or psychological disorder not related to shoulder instability compromising return to sports
4. Have a language barrier to complete the questionnaires in German
5. Are legally incapable of participating in research studies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2024-08-01 (Actual); Primary Completion 2025-05-31 (Actual); Study Completion 2025-05-31 (Actual)

PRIMARY OUTCOMES:
Shoulder Instability Return to Sports Index - German (SIRSI-D) | Baseline and after one week
  The SIRSI has been adapted to the shoulder instability cohort from the Anterior Cruciate Ligament Return to Sport Index (ACL-RSI) by (Gerometta et al., 2018). It is composed of twelve items that are rated on a zero to ten. The single total score is calculated by multiplying the sum of each item and dividing it by 120. The worst score then is zero indicating no psychological readiness to RTS and 100 the best, indicating full psychological readiness to RTS.
Tampa Scale for Kinesiophobia Shoulder Instability German (TSK-SI-D) | Baseline and after one week
  The TSK-SI has been adapted to the shoulder cohort by van Iersel et al (2023). The TSK-SI is composed of 18 questions scored on a 4 point Likert-Scale from "Strongly agree" to "Strongly disagree". The lowest score is 18, indicating no kinesiophobia and 72, indicating highest level of kinesiophobia.

SECONDARY OUTCOMES:
Western Ontario Shoulderinstability Index German (WOSI) | Baseline
  The the Western Ontario Shoulderinstability Index (WOSI) was developed by Kirkley (2003) and is the most prominent PROM in clinic and research for shoulder instability. The WOSI consists of 21 items and four domains: Physical symptoms (10 items), Sports, recreation, and work (4 items), lifestyle (4 items) and emotions (3 items). The scale for each item ranges from 0 to 100, allowing for a total score of 0 (best) to 2100 (worst).
SSV | Baseline
  The subjective shoulder value (SSV) was introduced by Gilbart and Gerber (2007) and provides a simple measure to represent shoulder functionality during activities of daily living (ADL). Patients are asked to rate their overall shoulder state on a scale from 0 to 100 percent, where a healthy shoulder is 100 percent. The scale results in a value between zero and 100, where zero means no subjective functionality during ADLs.
sSSV | Baseline
  Because the standard SSV might lack sport specific context Descamps et al (2023) suggested the sport subjective shoulder value (sSSV) with the question "Regarding sports practice, what is the overall percent value of your shoulder, if a completely normal shoulder represents 100% and a non-functional shoulder represents 0%?". The scale results in a value between zero and 100, where zero means no subjective functionality during sport.
Return to Sports Status | Baseline
  Ardern et al (2016) defined RTS as that the athlete has returned to his previous sport but not necessarily at the same performance level and differentiated it to return to participation and return to performance. This spectrum will be assessed using custom build questions to determine the RTS level

CONTACTS AND LOCATIONS:
Overall Officials: Asimina Lazaridou, PhD, Principal Investigator — Schulthess Klinik Zürich
Locations (1):
- Schulthess Klinik, Zurich, Switzerland

REFERENCES:
- [Background] van Iersel TP, Larsen van Gastel M, Versantvoort A, Hekman KMC, Sierevelt IN, Broekman BFP, van den Bekerom MPJ; Dutch Shoulder Instability Group (DSIG). The Modified Tampa-Scale of Kinesiophobia for Anterior Shoulder Instability. Arthrosc Sports Med Rehabil. 2023 Jul 24;5(4):100768. doi: 10.1016/j.asmr.2023.100768. eCollection 2023 Aug. PMID 37645388
- [Background] Gerometta A, Klouche S, Herman S, Lefevre N, Bohu Y. The Shoulder Instability-Return to Sport after Injury (SIRSI): a valid and reproducible scale to quantify psychological readiness to return to sport after traumatic shoulder instability. Knee Surg Sports Traumatol Arthrosc. 2018 Jan;26(1):203-211. doi: 10.1007/s00167-017-4645-0. Epub 2017 Jul 13. PMID 28707114

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-07-09): https://cdn.clinicaltrials.gov/large-docs/91/NCT06555991/Prot_SAP_001.pdf